CLINICAL TRIAL: NCT03684057
Title: Targeting Worry to Improve Sleep Using App-Based Mindfulness Training
Brief Title: Targeting Worry to Improve Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AG062004 (NIH); R21AG062004 (NIH)
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Anxiety; Sleep Disturbance
Keywords: Worry
MeSH Terms: conditions — Anxiety Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + App-Delivered Mindfulness Training (MT) (Experimental): The Unwinding Anxiety program is delivered via a smartphone-based platform, which includes a progression through 30+ daily modules of brief didactic and experience-based mindfulness training (videos and animations), app-triggered check-ins to encourage engagement, and user-initiated guided mindfulness exercises to help disrupt worry cycles in the moment.
  Interventions: Behavioral: App-Delivered Mindfulness Training (MT)
- Treatment as Usual (TAU) (Other): Individuals in the TAU group will complete the assessments without an intervention. (Note: participants will be transitioned to the Unwinding Anxiety program following the 2-month wait list control period)
  Interventions: Behavioral: App-Delivered Mindfulness Training (MT)

INTERVENTIONS:
Behavioral: App-Delivered Mindfulness Training (MT) — Unwinding Anxiety is an app-delivered mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on the self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time

SUMMARY:
The purpose of this study is to test an app-based mindfulness training program for worry to see if it can help individuals decrease worry and improve sleep.

DETAILED DESCRIPTION:
In this study, 80 individuals with worry interfering with sleep will be randomized to receive Unwinding Anxiety or to Treatment as Usual (50/50 chance). The active intervention period will last 2 months, with an optional 2-month follow-up period in which the intervention remains available. Changes in mindfulness, emotional reactivity, cognition and sleep behavior at specified time points will be measured. The primary engagement targets will be non-reactivity and worry. The primary behavioral outcome target will be sleep.

ELIGIBILITY:
Inclusion Criteria:

* Score > 40 on the Penn State Worry Questionnaire (PSWQ)
* Score ≥ to 40% on Worry Interfering with Sleep Scale (WISS)
* Owns a smartphone
* Willing to wear a sleep tracker for at least 1 week

Exclusion Criteria:

* Any usage of psychotropic medication: not on a stable dosage 6+ weeks
* Medical disorder of the severity that would interfere with ability to attend visits and complete study milestones
* Use of benzodiazepine or hypnotic sleep aid on as needed (i.e. prn)
* Known sleep disorder
* Psychotic disorder
* Post-traumatic Stress Disorder
* Severe depression (Score > 3 on PHQ-2)
* Current shift work employment
* BMI > 35
* Evening caffeine use
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judson Brewer, MD, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao M, Roy A, Deluty A, Sharkey KM, Hoge EA, Liu T, Brewer JA. Targeting Anxiety to Improve Sleep Disturbance: A Randomized Clinical Trial of App-Based Mindfulness Training. Psychosom Med. 2022 Jun 1;84(5):632-642. doi: 10.1097/PSY.0000000000001083. Epub 2022 Apr 14. PMID 35420589

RESULTS

PARTICIPANT FLOW:
Groups:
- TAU and App-delivered Mindfulness Training (MT): Unwinding Anxiety is an app-delivered mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on the self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time
- Treatment as Usual (TAU): Individuals in the TAU group will complete the assessments without an intervention. (Note: participants will be transitioned to the Unwinding Anxiety program following the 2-month wait list control period)
  App-based mindfulness training: Unwinding Anxiety is an app-based mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on the self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time
Period: Overall Study
Arm/Group | TAU and App-delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
Started | 40 | 40
Completed | 36 | 35
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Population: The 4 participants in the TAU group and 5 participants in the TAU + MT group who withdrew from the study were excluded from analyses.
Groups:
- TAU + App-Delivered Mindfulness Training (MT): Unwinding Anxiety is an app-delivered mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on the self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time
- Total: Total of all reporting groups
Arm/Group | TAU + App-Delivered Mindfulness Training (MT) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (18.5) | 40.6 (16.8) | 41 (18)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 9 | 3 | 12
  Female | 25 | 32 | 57
  Prefer not to answer | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 23 | 44
  Black/African American | 1 | 0 | 1
  Hispanic, Latinx, Spanish | 2 | 3 | 5
  Asian | 6 | 5 | 11
  ≥2 races | 6 | 4 | 10
Highest level of education completed [Count of Participants; unit: Participants]
  High school or GED | 2 | 0 | 2
  Some college | 4 | 8 | 12
  Associate's degree | 2 | 3 | 5
  Bachelor's degree | 11 | 8 | 19
  Graduate degree | 17 | 16 | 33
Work status [Count of Participants; unit: Participants]
  Employed full-time | 19 | 22 | 41
  Employed part-time | 12 | 6 | 18
  Homemaker | 1 | 0 | 1
  Retired | 2 | 3 | 5
  Unemployed | 2 | 4 | 6
Marital status [Count of Participants; unit: Participants]
  Never married | 17 | 16 | 33
  Married | 9 | 16 | 25
  Separated/divorced | 7 | 2 | 9
  Widowed | 3 | 1 | 4
Income [Count of Participants; unit: Participants]
  <$15,000-$44,999 | 9 | 6 | 15
  $45,000-$99,999 | 12 | 9 | 21
  ≥$100,000 | 12 | 10 | 22
  Prefer not to answer | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Worry-related Sleep Disturbances
Description: 5 questions from the 29-item Patient-Reported Outcomes Measurement Information System (PROMIS-29) pertaining to anxiety and sleep will be used to assess worry-related sleep disturbances over the past 7 days. These questions are on a 5-point Likert scale where 1 is "Not at all" and 5 is "Very much". Scores can range from 5 to 25 and higher scores indicate a worse outcome.
Time Frame: Baseline, 2 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAU + App-Delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 35
units on a scale | -4 [-8.0 to -2.8] | -1 [-4 to 2.0]

2. Secondary Outcome: Change in Worry
Description: Penn State Worry Questionnaire (PSWQ) will be used to assess worry. The PSWQ is a 16-item questionnaire that uses a 5-point Likert scale where 1 is "Not at all typical of me" and 5 is "Very typical of me". Scores can range from 16 to 80 and higher scores indicate a worse outcome
Time Frame: Baseline, 2 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAU and App-delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 35
units on a scale | -9 [-12.2 to -1.0] | 0.0 [-4.0 to 2.5]

3. Secondary Outcome: Change in Total Sleep Time (TST)
Description: A Fitbit will be used to assess sleep trends over a 1 week period
Time Frame: Baseline, 2 months
Population: Fitbit data was not available for both wear periods (due to a failure to wear and/or technical issues) for 11 participants in the TAU + MT group and for 14 participants in the TAU group.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | TAU and App-delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 25 | 21
minutes | 9 [-28 to 34] | 3 [-21 to 37]

4. Secondary Outcome: Changes in Non-reactivity
Description: Non-reactivity subscale from the 15-item Five Facet Mindfulness Questionnaire (FFMQ) will be used to measure changes in emotional reactivity. This subscale is based on responses to 3 questions measured on a 5-point Likert scale where 1 is "Never or rarely" and 5 is "Very often or always true". Scores can range from 3 to 15 and higher scores indicate a better outcome.
Time Frame: Baseline, 2 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAU + App-Delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 35
units on a scale | 4.5 [1.0 to 6.0] | 0 [-2.0 to 2.5]

ADVERSE EVENTS:
Time Frame: 4 months
Description: All participants were assessed for adverse events at their final study visit (conclusion of study).
Arm/Group | TAU and App-delivered Mindfulness Training (MT) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03684057/Prot_SAP_001.pdf
  • Informed Consent Form (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03684057/ICF_000.pdf